CLINICAL TRIAL: NCT07017400
Title: Effectiveness of the Sacral Erector Spinae Plane (ESP) Block in Total Knee Arthroplasty: A Prospective Observational Study
Brief Title: The Sacral Erector Spinae Plane Block in Total Knee Arthroplasty
Acronym: sacral ESP
Status: Recruiting | Type: Observational
Sponsor: San Giovanni di Dio Hospital (Other)
Responsible Party: Principal Investigator, Tommaso Sorrentino, Principal Investigator, San Giovanni di Dio Hospital
Other Study IDs: 143/2025
Record Dates: First submitted 2025-05-24; First posted 2025-06-12 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Total Knee Anthroplasty; Regional Anesthesia
Keywords: regional anesthesia; total knee arthroplasty
MeSH Terms: interventions — Anesthetics, Local

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACB/iPACK: combination of adductor canal block (saphenous) and infiltration between the Popliteal Artery and Capsule of the Knee (iPACK) block
  Interventions: Procedure: Local Anesthetic Injection
- ACB/sacral ESP: combination of adductor canal block (saphenous) and sacral erector spinae plane (ESP) block
  Interventions: Procedure: Local Anesthetic Injection

INTERVENTIONS:
Procedure: Local Anesthetic Injection — combination of regional blocks for TKA postoperative analgesia

SUMMARY:
The goal of this observational study is to learn about the analgesic efficacy and postoperative recovery of two locoregional anesthesia combinations in patients > 18 years (ASA I-III), scheduled for unilateral TKA under spinal anesthesia with expected hospitalization > 24 hours:

* ACB + sacral ESP block
* ACB + iPACK block

The main question it aims to answer is: Does the ACB + sacral ESP block combination produce effective postoperative recovery and analgesic effect?

Participants already taking ACB + sacral ESP block as part of their regular peri-operative care for TKA will be followed in the postoperative period for 48 hours.

DETAILED DESCRIPTION:
Total Knee Arthroplasty (TKA) is a common orthopedic surgery in elderly patients, often requiring effective postoperative pain control to enhance recovery. Conventional locoregional techniques include adductor canal block (ACB) and the iPACK block (infiltration between the Popliteal Artery and Capsule of the Knee). While effective, iPACK may carry infection risks due to its proximity to the surgical field.

The sacral ESP block is a more recent ultrasound-guided technique targeting posterior sacral nerve branches from a remote site, potentially avoiding motor weakness and surgical site complications. Early literature and local clinical experience suggest that combining sacral ESP with ACB may provide comparable analgesia to ACB+iPACK while offering practical and safety advantages.

Study Design:

* Type: Single-center, prospective, observational study
* Setting: Ospedale di Crotone, Italy
* Duration: Maximum of 30 months
* Sample size: 63 patients per group (based on QoR-15 score, with 80% power and α = 0.05)

Population:

* Adults >18 years (ASA I-III), scheduled for unilateral TKA with expected hospitalization >24 hours
* Exclusion: refusal of consent, contraindications to spinal or regional anesthesia, coagulation disorders, severe dementia, ongoing infection, or emergency surgeries

Primary Endpoint:

* Quality of Recovery (QoR-15) score at 24 hours post-surgery (score range 0-150; higher scores indicate better recovery)

Secondary Endpoints:

* Postoperative pain scores (NRS, score range 0-10, higher scores indicate more pain) at rest and movement (0-48 hours)
* Time to first mobilization
* Patient satisfaction (Likert scale)
* Analgesic consumption and time to first request
* Incidence of nausea, vomiting, antiemetic use
* Block-related complications or adverse events

Procedure:

All patients receive spinal anesthesia and multimodal postoperative analgesia (paracetamol, rescue tramadol). Regional blocks are performed under ultrasound guidance in aseptic conditions. ESP is performed at the S2 level with 20 mL ropivacaine 0.375%. ACB and iPACK are also administered per standard protocols.

Data Analysis:

Statistical comparisons between groups will be made using appropriate parametric or non-parametric tests based on variable distribution. Repeated measures will be analyzed using linear mixed-effects models.

Ethics:

The study follows Good Clinical Practice (GCP) and the Declaration of Helsinki. Patients provide written informed consent. Privacy and data confidentiality are ensured.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years
* ASA I-III
* scheduled for unilateral TKA with expected hospitalization > 24 hours

Exclusion Criteria:

* Refusal of consent
* Local anesthetics allergies
* contraindications to spinal or regional anesthesia
* coagulation disorders
* anticoagulation/antiaggregation medications
* dementia
* ASA-PS > III
* ongoing infection
* emergency surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults >18 years scheduled for unilateral TKA
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery (QoR-15) score at 24 hours post-surgery | at 24 hours post-surgery
  Quality of Recovery (QoR-15) - score range 0-150 - higher scores indicate better recovery

SECONDARY OUTCOMES:
Postoperative pain scores (NRS) at rest and movement (0-48 hours) | 0-48 hours from surgery
  NRS at rest and movement - score range 0 (no pain) - 10 (the worst pain)
Time to first mobilization | 0-48 hours
  first patient mobilization - time (hour) of first mobilization
Analgesic consumption (total drug dosage) | 0-48 hours
  Effectiveness of the blocks
Time to first analgesic request (time - hour - of first request) | 0-48 hours
  Duration of the blocks

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni Crotone Hospital, Crotone, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marrone F, Fusco P, Paventi S, Pullano C. Combined adductor canal (ACB) and sacral erector spinae plane (S-ESP) blocks for total knee arthroplasty pain in hemophilic arthropathy. Saudi J Anaesth. 2024 Oct-Dec;18(4):565-568. doi: 10.4103/sja.sja_177_24. Epub 2024 Oct 2. PMID 39600436
- [Background] Marrone F, Pullano C, Paventi S, Tomei M, Fusco P. A unilateral single level sacral erector spinae plane block for total knee arthroplasty pain. Minerva Anestesiol. 2024 Jul-Aug;90(7-8):707-708. doi: 10.23736/S0375-9393.24.18046-7. Epub 2024 Feb 29. No abstract available. PMID 38421355
- [Background] Marrone F, Fusco P, Paventi S, Tomei M, Lolli S, Chironna E, Pullano C. Combined lumbar and sacral erector spinae plane (LS-ESP) block for hip fracture pain and surgery. Minerva Anestesiol. 2024 Jul-Aug;90(7-8):712-714. doi: 10.23736/S0375-9393.24.18093-5. Epub 2024 Apr 24. No abstract available. PMID 38656087
- [Background] Marrone F, Paventi S, Tomei M, Failli S, Crecco S, Pullano C. Unilateral sacral erector spinae plane block for hip fracture surgery. Anaesth Rep. 2024 Jan 3;12(1):e12269. doi: 10.1002/anr3.12269. eCollection 2024 Jan-Jun. PMID 38187935
- [Background] Satici MH, Tutar MS, Tire Y, Binici O, Cicekler O, Korkmaz E, Pekince O, Kozanhan B. The effect of sacral erector spinae plane block on the quality of recovery after total hip arthroplasty: a prospective, randomized, controlled, multicenter study. Minerva Anestesiol. 2025 Apr;91(4):278-285. doi: 10.23736/S0375-9393.24.18353-8. Epub 2024 Nov 4. PMID 39495168
- [Background] Tulgar S, Senturk O, Thomas DT, Deveci U, Ozer Z. A new technique for sensory blockage of posterior branches of sacral nerves: Ultrasound guided sacral erector spinae plane block. J Clin Anesth. 2019 Nov;57:129-130. doi: 10.1016/j.jclinane.2019.04.014. Epub 2019 Apr 15. No abstract available. PMID 30999197
- [Background] Lavand'homme PM, Kehlet H, Rawal N, Joshi GP; PROSPECT Working Group of the European Society of Regional Anaesthesia and Pain Therapy (ESRA). Pain management after total knee arthroplasty: PROcedure SPEcific Postoperative Pain ManagemenT recommendations. Eur J Anaesthesiol. 2022 Sep 1;39(9):743-757. doi: 10.1097/EJA.0000000000001691. Epub 2022 Jul 20. PMID 35852550